CLINICAL TRIAL: NCT04626284
Title: Clinical Trial to Evaluate the Safety and Effectiveness of Normothermic Regional Perfusion (NRP) for Resuscitation of Hearts From Donation After Circulatory Death (DCD)
Brief Title: Safety and Effectiveness of NRP for DCD Heart Transplantation
Acronym: DCDNRPHeart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0460-20-FB
Record Dates: First submitted 2020-11-02; First posted 2020-11-12 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Heart Transplant Failure; Determination of Death; Outcomes Research; Death
Keywords: Heart transplantation; Donation after circulatory death; Normothermic regional perfusion
MeSH Terms: conditions — Death | interventions — Heart Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donors After Circulatory Determined death (Experimental): Recipients receiving an organ from donors after circulatory determined death
  Interventions: Procedure: Heart Transplantation

INTERVENTIONS:
Procedure: Heart Transplantation — Heart Transplantation

SUMMARY:
This is a prospective, observational, pilot trial to evaluate the feasibility of heart transplantation using normothermic regional perfusion (NRP) donation after donor circulatory death (DCD). Normothermic regional perfusion utilizes Extracorporeal Membrane Oxygenation (ECMO) or cardiopulmonary bypass to reperfuse the heart and other organs in situ after isolation and ligation of the cerebral vessels. In situ resuscitation of the heart has the added advantage of allowing full hemodynamic and echocardiographic assessment of the donor heart prior to final acceptance for transplantation without the imminent danger of ongoing warm ischemia.

DETAILED DESCRIPTION:
The current procedure of DCD organ donation and procurement follows a well-established course for lung, liver, kidney and pancreas transplantation in the United States. DCD transplantation of a heart has been hampered due to concern about the graft viability after the obligatory period of warm ischemia and also the limited ability to assess the graft function after the cessation of circulation. Normothermic regional perfusion restores the circulation and enables in-situ reanimation of thoracic and abdominal organs after the circulatory determination of death. For heart transplantation, the investigators will accept donors between the ages of 18 and 49 without any known history of coronary artery disease, insulin dependent diabetes, or long-term smoking (>20 pack/years) and normal baseline cardiac function (EF>50) assessed with transthoracic echocardiogram. After the authorization for research has been obtained from DCD surrogate, the organs will be allocated through UNOS. When all parties are present and ready, the donor will be withdrawn from life support (i.e., discontinuation of mechanical ventilation and any vasoactive medications). . After circulatory arrest occurs, death is declared by a physician not associated with the transplant teams. Subsequently a period of stand-off is observed (5 minutes for organs donated in Nebraska) to ensure complete cessation of the circulation before organ procurement is commenced. If after withdrawal of life support the patient does not progress to circulatory death within the allotted time, the procurement is abandoned and the patient is transferred out of the operating room and placed on palliative measures.

Given that DCD organ donation is already currently practiced in the US, the same standard approach defined by each state and locality can also be applied to DCD heart donation and will be followed for this protocol at UNMC. However, this protocol will utilize a normothermic regional perfusion (NRP) strategy that involves reestablishment of circulatory blood flow after the period of circulatory arrest has been established and the 5 minutes of standoff time has passed. The local Organ Procurement Organization (LiveOnNE) have reviewed and approved this approach to DCD heart donation. Specifically, normothermic regional perfusion involves the following steps:

1. Opening the chest through a standard sternotomy used for heart and lung procurement.
2. Ligation of the all the blood vessels that supply blood to the brain to ensure that blood flow to the brain is not reestablished once circulation is restarted as described below.
3. Standard cannulation of the aorta and the right atrium as is done for cardiac surgical procedures.
4. Initiation of cardiopulmonary bypass, which will re-establish the flow of blood to all organs of the body including the heart under normothermia. The initial step for ligation of the blood vessels to the head is necessary to ensure that blood flow to the brain does not occur.

Once blood flow to the heart is established, the heart will start beating. At 30 minute intervals, the donor will be separated from cardiopulmonary bypass and the heart will be assessed for functionality. If accepted standard DBD procurement will commence. The heart transplantation surgery on the potential recipient will only begin once the heart has been accepted as suitable.

If after assessment the heart is not suitable, cardiopulmonary bypass will be restarted. The donor heart will be reassessed at 30-minute intervals up to 180 minutes. If no significant acceptable recovery occurs and the heart is not deemed suitable for transplantation, then the study will be terminated, but the remaining organs can be recovered as standard practice.

ELIGIBILITY:
Inclusion Criteria:

1. Recipient is ≥ 19 years old
2. Recipient, or their designated healthcare proxy, is able and willing to sign informed consent
3. Recipient meets standard listing criteria for heart transplantation

Exclusion Criteria:

1. Recipient is < 19 years old
2. Recipient, or their designated healthcare proxy, is unable to sign informed consent
3. Recipient is participating in another interventional trial
4. Recipient has a known history of HIV infection
5. Recipient has any condition that, in the opinion of the Investigator, would make study participation unsafe or would interfere with the objectives of the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Utilization rate | Date from the first DCD NRP Heart procurement until the 25th DCD NRP heart procurement, assessed up to 36 months
  Ratio of successful heart transplants using grafts obtained from DCD donors using NRO to the total number of DCD donors in whom NRP was used to procure an organ

SECONDARY OUTCOMES:
Graft survival | From date of the transplantation to date of death or retransplantation, whichever comes first, assessed up to 12 months
  Survival of the graft censored either at the time of death of the recipient or retranaplantation
Primary Graft Dysfunction (PGD) | From day of heart transplantation up to 72 hours post-transplantation
  Primary Graft Dysfunction as defined by ISHLT
Acute cellular rejection (ACR) | From day of heart transplantation up to 1 year post-transplantation
  Biopsy proven acute cellular rejection requiring treatment
Antibody mediated rejection (AMR) | From day of heart transplantation up to 1 year post-transplantation
  Biopsy proven antibody mediated rejection

CONTACTS AND LOCATIONS:
Overall Officials: Marian Urban, MD, PhD, Principal Investigator — Assistant Professor
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barnard CN. The operation. A human cardiac transplant: an interim report of a successful operation performed at Groote Schuur Hospital, Cape Town. S Afr Med J. 1967 Dec 30;41(48):1271-4. No abstract available. PMID 4170370
- [Result] Dhital KK, Chew HC, Macdonald PS. Donation after circulatory death heart transplantation. Curr Opin Organ Transplant. 2017 Jun;22(3):189-197. doi: 10.1097/MOT.0000000000000419. PMID 28379853
- [Result] Messer S, Page A, Colah S, Axell R, Parizkova B, Tsui S, Large S. Human heart transplantation from donation after circulatory-determined death donors using normothermic regional perfusion and cold storage. J Heart Lung Transplant. 2018 Jul;37(7):865-869. doi: 10.1016/j.healun.2018.03.017. Epub 2018 Mar 30. PMID 29731238
- [Result] Chew HC, Iyer A, Connellan M, Scheuer S, Villanueva J, Gao L, Hicks M, Harkness M, Soto C, Dinale A, Nair P, Watson A, Granger E, Jansz P, Muthiah K, Jabbour A, Kotlyar E, Keogh A, Hayward C, Graham R, Spratt P, Macdonald P, Dhital K. Outcomes of Donation After Circulatory Death Heart Transplantation in Australia. J Am Coll Cardiol. 2019 Apr 2;73(12):1447-1459. doi: 10.1016/j.jacc.2018.12.067. PMID 30922476